CLINICAL TRIAL: NCT01100827
Title: A Retrospective Molecular Epidemiology Study in Singapore Patients With Advanced Non Small Cell Lung Cancer (NSCLC) of Adenocarcinoma Histology to Assess Epidermal Growth Factor Receptor (EGFR) Mutation Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: NS01/03/10
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: NSCLC
Keywords: EGFR mutation status in patients with advanced stage adenocarcinoma NSCLC; The association between EGFR mutation status and demographic data in advanced stage adenocarcinoma NSCLC patients.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- EGFR mutation status in patients
  Interventions: Other: EGFR mutation status in patients

INTERVENTIONS:
Other: EGFR mutation status in patients

SUMMARY:
To determine EGFR mutation status in patients with advanced stage adenocarcinoma NSCLC.

To determine the association between EGFR mutation status and demographic data in advanced stage adenocarcinoma NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

Nil

Exclusion Criteria:

Nil

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In order to determine the EGFR mutation status, data analysis will be performed on demographic data and medical records (i.e. case notes and pathology reports) from patient with advanced stage adenocarcinoma NSCLC
Sampling Method: Probability Sample
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital Singapore, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Shigematsu H, Lin L, Takahashi T, Nomura M, Suzuki M, Wistuba II, Fong KM, Lee H, Toyooka S, Shimizu N, Fujisawa T, Feng Z, Roth JA, Herz J, Minna JD, Gazdar AF. Clinical and biological features associated with epidermal growth factor receptor gene mutations in lung cancers. J Natl Cancer Inst. 2005 Mar 2;97(5):339-46. doi: 10.1093/jnci/dji055. PMID 15741570
- [Background] Miller VA, Kris MG, Shah N, Patel J, Azzoli C, Gomez J, Krug LM, Pao W, Rizvi N, Pizzo B, Tyson L, Venkatraman E, Ben-Porat L, Memoli N, Zakowski M, Rusch V, Heelan RT. Bronchioloalveolar pathologic subtype and smoking history predict sensitivity to gefitinib in advanced non-small-cell lung cancer. J Clin Oncol. 2004 Mar 15;22(6):1103-9. doi: 10.1200/JCO.2004.08.158. PMID 15020612